CLINICAL TRIAL: NCT06286787
Title: Efficacy of Mountain Craft Training at Enhancing the Resilience and Physical and Psychological Well-being of Children From Low-income Families: A Pilot Randomised Controlled Trial
Brief Title: Efficacy of Mountain Craft Training at Enhancing the Resilience and Physio-psychological Well-being of Children From Low-income Families
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Joyce Chung, Assistant Professor, School of Nursing, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSEARS20221110002
Record Dates: First submitted 2024-02-15; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Resilience; Well-being; Children
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in the intervention group will be invited to join the mountain craft training programme.
  Interventions: Other: Intervention
- Placebo control group (Placebo Comparator): Participants will be invited to join a control intervention that mimics the time and attention received by participants in the intervention group but will be designed to have no specific effect on the outcome variables.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Intervention — The training programme will consist of a 3-hour lecture. The contents of the lecture will include knowledge of mountaineering in Hong Kong, country codes and care for the environment, environmental awareness when undertaking outdoor activities, hiking skills, knowledge and choice of hiking equipment and clothing, trip planning, mountain safety, map reading, the use of a compass, mountain safety, basic first aid, methods of calling for help in an emergency and sources of weather data. After completing the lecture, participants will be required to join a 6-day hiking training programme on weekends within a 3-month period (each training will be at least 5 kilometres and the duration will be at least 4 hours).
  Arms: Intervention group
Other: Placebo — Control participants will be asked to join six day-time leisure activities on weekends within a 3-month period. Leisure activities will be organised by the Asbury Methodist Social Service and will include cartoon film shows, handicraft workshops, chess games, health talks on the prevention of influenza and eating a healthy diet, and day visits to a museum and theme park. Children in the placebo control group will receive free access to leisure activities, including visits to museums and theme parks as an incentive for his/her participation.
  Arms: Placebo control group

SUMMARY:
It is imperative to offer adequate community resources and psychosocial support, with a particular focus on enhancing resilience for children from low-income families. This study aims to determine the feasibility, acceptability, and preliminary efficacy of mountain craft training in enhancing resilience and self-esteem, reducing depressive symptoms, and improving the physical health of children from low-income families.

DETAILED DESCRIPTION:
It is imperative to offer adequate community resources and psychosocial support, with a particular focus on enhancing resilience for children from low-income families. This study aims to determine the feasibility, acceptability, and preliminary efficacy of mountain craft training in enhancing resilience and self-esteem, reducing depressive symptoms, and improving the physical health of children from low-income families. This will be a pilot RCT using a two-group pre- and post-test within-subject design. The investigators plan to recruit 40 children in the Kwai Tsing District to participate in this study via the Asbury Methodist Social Service. Participants in the intervention group will be invited to join the mountain craft training programme. The research team will work with Mountain & Stream (https://www.mtandstream.com/) to offer a tailor-made hiking training programme for Form 1 students. Participants will be invited to join a control intervention that mimics the time and attention received by participants in the intervention group but will be designed to have no specific effect on the outcome variables. The investigators hypothesise that participants who receive mountain craft training (six sessions) over 3 months will report significant improvements in: (i) resilience, (ii) self-esteem; (iii) depressive symptoms, and (iv) physical well-being compared with those in the placebo control group at the 6-month follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Form 1 students
* able to speak Cantonese and read Chinese, and
* from low-income families (with a half-median monthly household income or the recipients of Comprehensive Social Security Assistance)

Exclusion Criteria:

* Children with identified cognitive or learning problems, chronic illness, or physical disabilities

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Resilience Scale-14 (RS-14) | baseline, 3-month, and 6-month
  The RS-14 will be used to measure participants' resilience. The RS-14 measures two factors: personal competence and acceptance of self and life.24 Each item is answered on a 7-point Likert scale from 'strongly disagree' to 'strongly agree', with total scores ranging from 14 to 98. Higher scores indicate higher levels of resilience. The RS-14 has been translated into Chinese and used to measure children's resilience in a previous study.25 The psychometric properties of the Chinese version of the RS-14 have been tested, with a test-retest reliability of .84 and internal consistency (Cronbach's α) of .86.

SECONDARY OUTCOMES:
Chinese version of the Center for Epidemiologic Studies Depression Scale for Children (CES-DC) | baseline, 3-month, and 6-month
  Participants' depressive symptoms will be evaluated using the CES-DC, which contains 20 completely standardized items to assess depressive symptoms. All items are scored on a 4-point self-report scale ranging from 0 to 3 corresponding to their occurrence in the previous week. Total scores range from 0 to 60, with higher scores indicating more prominent symptomatology. The psychometric properties of the Chinese version of the CES-DC have been tested; the version has a high content legitimacy (content legitimacy index = 95%) and satisfactory internal consistency reliability (r = 0.82).
Chinese version of Rosenberg's Self-Esteem Scale (RSES) | baseline, 3-month, and 6-month
  Participants' self-esteem will be evaluated using the RSES, which contains includes 10 items intended to evaluate the self-esteem of children and adolescents worldwide. Each item is scored on a 4-point Likert scale ranging from 1 to 4, with total scores ranging from 10 to 40. Higher scores demonstrate higher levels of self-esteem. The Chinese version of the RSES has recently been used in Chinese children, and has shown sufficient internal reliability (r = 0.84).
The children's peak expiratory flow rate | baseline, 3-month, and 6-month
  A miniWright Standard Handheld peak flow meter will be used for measuring peak expiratory flow rate.

CONTACTS AND LOCATIONS:
Locations (1):
- The Asbury Methodist Social Service, Hong Kong, China